CLINICAL TRIAL: NCT06111404
Title: Lateral Versus Central Urinary Bladder Dissection During Total Laparoscopic Hysterectomy in Cases With Previous Cesarean Section: A Randomized Controlled Study
Brief Title: Urinary Bladder Dissection During Total Laparoscopic Hysterectomy in Cases With Previous Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD.22.11.720
Record Dates: First submitted 2023-10-03; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Total Laparoscopic Hysterectomy
Keywords: urinary bladder dissection; total laparoscopic hysterectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (central group) (Active Comparator): A metal catheter was then inserted in the bladder. The catheter was rotated so the tip was pointing upward, to stretch the bladder pillars. The bladder was dissected with monopolar scissors with the catheter in place. Then opening the posterior leaflet of the broad ligament to the cervix, opening of the vesico-vaginal space and dissecting the bladder downwards will be done (Poojari et al., 2014). Coagulation and section of the uterine pedicles: performed on the ascending segment of the uterine artery, will be carried out in a progressive manner on both sides.
  Interventions: Procedure: central urinary bladder dissection; Device: Wolf laparoscopy tower
- Group B (lateral group) (Active Comparator): The broad ligament is dissected down till the uterine bundle is identified. Once the uterine vascular bundle is identified the space can be dissected just above these vessels to reach the lateral margins of cervix. Any fatty tissue should be moved with the bladder. Uterine vessels are then tackled by desiccation or ligation. Similar procedure is done on the opposite side. Once the bladder is completely dissected and lifted off from the cervix below, midline adhesions of the bladder and pillars can be gradually separated using sharp dissection or Ligasure staying near to cervix (Chen et al., 2007).
  Interventions: Procedure: Lateral urinary bladder dissection; Device: Wolf laparoscopy tower

INTERVENTIONS:
Procedure: central urinary bladder dissection — A metal catheter was then inserted in the bladder. The catheter was rotated so the tip was pointing upward, to stretch the bladder pillars. The bladder was dissected with monopolar scissors with the catheter in place. Then opening the posterior leaflet of the broad ligament to the cervix, opening of the vesico-vaginal space and dissecting the bladder downwards will be done (Poojari et al., 2014). Coagulation and section of the uterine pedicles: performed on the ascending segment of the uterine artery, will be carried out in a progressive manner on both sides.
  Arms: Group A (central group)
Procedure: Lateral urinary bladder dissection — The broad ligament is dissected down till the uterine bundle is identified. Once the uterine vascular bundle is identified the space can be dissected just above these vessels to reach the lateral margins of cervix. Any fatty tissue should be moved with the bladder. Uterine vessels are then tackled by desiccation or ligation. Similar procedure is done on the opposite side. Once the bladder is completely dissected and lifted off from the cervix below, midline adhesions of the bladder and pillars can be gradually separated using sharp dissection or Ligasure staying near to cervix (Chen et al., 2007).
  Arms: Group B (lateral group)
Device: Wolf laparoscopy tower — set of instruments used for laparoscopic surgery

SUMMARY:
Mobilization of the urinary bladder off of the cervix is an important step in total laparoscopic hysterectomy, and is always performed before dealing with the uterine pedicle. If the uterus is unscarred, bladder mobilization may not be technically difficult. However, if the uterus is scarred, there can be adhesions not only between the uterus and the bladder but also to the anterior abdominal wall, which can make dissection challenging. Studies of the effects of closure or nonclosure of the peritoneum during cesarean delivery on adhesion formation have concluded that insufficient data are available and that adequately powered and designed trials are needed.

As regards the lateral approach, this space was first described by Dr. Shrish Sheth utilizing the utero-cervical broad ligament in post cesarean cases during vaginal hysterectomy. He described that the lateral area; the two leaves of broad ligament remains free and allows easy possibility for entry to dissect whether vaginally or abdominally. While in medial approach, a metal catheter was then inserted in the bladder. The catheter was rotated so the tip was pointing upward, to stretch the bladder pillars. The bladder was dissected with monopolar scissors with the catheter in place.

DETAILED DESCRIPTION:
Hysterectomy is one of the most commonly performed gynecological operations. It is carried out because of a variety of indications, such as presence of dysfunctional uterine bleeding, myoma uteri, adenomyosis and adnexal mass. Hysterectomy can be performed using abdominal, vaginal, laparoscopic or robotic methods. According to the results from a study performed in the United States, the incidence rates for hysterectomies using abdominal, vaginal and laparoscopic methods are 66%, 22% and 12%, respectively.

There is still no consensus on which of these approaches is the optimum surgical method for hysterectomy. Abdominal hysterectomy is the most frequently performed approach, but current clinical practice mandates that, when appropriate, the surgical method should be vaginal rather than abdominal, since the former is associated with better outcomes and lower complication rates. Moreover, when vaginal hysterectomy is not feasible or not indicated, the surgical method should be laparoscopic, because total laparoscopic hysterectomy (TLH) provides a faster return to normal activity, shorter hospital stays, lower intraoperative bleeding and fewer wound infections, compared with abdominal hysterectomy. However, longer operating times and higher incidence of urinary system damage are seen in laparoscopic hysterectomies.

Cesarean section (CS) is the most commonly performed surgery on women and has increased significantly in the last 15 years. Various reasons account for the increase in CS, including an increase upon maternal request, changes in maternal demographics (e.g., increasing maternal age), changes in physician practice patterns, more conservative practice guidelines, and mounting legal pressures.

Because of the gradually increasing rates of cesarean sections (CSs) over the last two decades, the number of hysterectomized patients with previous CS has increased. In a recent review article, previously performed CSs were demonstrated to be an important risk factor for lower urinary tract injuries, and the recommendation that abdominal hysterectomy might be preferable for these patients was emphasized. TLH may be technically difficult in patients with previous CSs, due to surgical adhesions, and is associated with a higher risk of perioperative complications.

Mobilization of the urinary bladder off of the cervix is an important step in total laparoscopic hysterectomy, and is always performed before dealing with the uterine pedicle. If the uterus is unscarred, bladder mobilization may not be technically difficult. However, if the uterus is scarred, there can be adhesions not only between the uterus and the bladder but also to the anterior abdominal wall, which can make dissection challenging. Studies of the effects of closure or nonclosure of the peritoneum during cesarean delivery on adhesion formation have concluded that insufficient data are available and that adequately powered and designed trials are needed.

As regards the lateral approach, this space was first described by Dr. Shrish Sheth utilizing the utero-cervical broad ligament in post cesarean cases during vaginal hysterectomy. He described that the lateral area; the two leaves of broad ligament remains free and allows easy possibility for entry to dissect whether vaginally or abdominally.While in medial approach, a metal catheter was then inserted in the bladder. The catheter was rotated so the tip was pointing upward, to stretch the bladder pillars. The bladder was dissected with monopolar scissors with the catheter in place.

ELIGIBILITY:
Inclusion Criteria:

.Patients undergoing total laparoscopic hysterectomy for benign conditions (e.g., dysfunctional uterine bleeding, adenomyosis and uterine fibroids) with presence of previous cesarean section scar.

Exclusion Criteria:

* Patients with prior abdominal surgery other than CS.
* Patients treated with concomitant surgery, including laparoscopic pelvic lymphadenectomy, posterior vaginal colporrhaphy and tension-free vaginal or obturator tape procedures.
* Tubo-ovarian abscess.
* Endometriosis.
* Pelvic tuberculosis.
* Pelvic organ prolapses. .Patients with relative contraindication to general anesthesia (e.g. chronic liver cell failure.

.Patients with contraindication to laparoscopic surgery (e.g. severe cardio-pulmonary dysfunction).

* Bleeding tendency (e.g. anticoagulants, platelets disorders)
* Body mass index more than 35 Kg/m2

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-22 (Actual); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the procedure | during urinary bladder dissection intraoperative
  rate of urinary bladder injury during dissection

SECONDARY OUTCOMES:
operative time | from time of primary port insertion till vault closure
  time of primary port insertion till vault closure
amount of blood loss | during whole procedure
  total blood loss in vacuum during surgery
late urological complications | intraoperative up to 2 months postoperative
  genitourinary fistula and ureteric injury

CONTACTS AND LOCATIONS:
Overall Officials: ahmed elawady, M.Sc, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
arms.inclusion and exclusion criteria